CLINICAL TRIAL: NCT02485613
Title: Bortezomib With Dexamethasone as the First-line Treatment for Immunoglobulin Light Chain(AL) Amyloidosis
Brief Title: Bortezomib for Immunoglobulin Light Chain(AL) Amyloidosis
Status: Completed | Type: Observational
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Other Study IDs: NJCT-1501
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Dexamethasone; Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bortezominb and dexamethasone group
  Interventions: Drug: bortezominb and dexamethasone

INTERVENTIONS:
Drug: bortezominb and dexamethasone — The initial BD regimen included bortezomib (1.3 mg/m2 i.v.) and dexamethasone (40 mg i.v.) twice weekly for 2 weeks (days 1, 4, 8, and 11), which was followed by a 10-day rest period (days 12-21). The dose of bortezomib and dexamethasone can be adjusted according to the patients' condition.
  Other Names: Velcade

SUMMARY:
Although the use of bortezomib has reported efficacy in amyloid light chain (AL) amyloidosis, the role of bortezomib with dexamethasone (BD) in the first-line treatment of patients with AL amyloidosis should be determined. In this study, the investigators evaluated the efficacy and safety of BD as the first-line treatment of patients with AL amyloidosis.

DETAILED DESCRIPTION:
This study included patients with newly diagnosed AL amyloidosis who were treated with a BD regimen in Jinling hospital. The AL amyloidosis diagnosis was confirmed by renal biopsy, and the assessment of organ involvement were based on consensus criteria. The clinical and laboratory data were collected at the beginning of each cycle and every 3 months thereafter. The initial BD regimen included bortezomib (1.3 mg/m2 i.v.) and dexamethasone (40 mg i.v.) twice weekly for 2 weeks (days 1, 4, 8, and 11), which was followed by a 10-day rest period (days 12-21). The investigators evaluated the efficacy and safety of BD as the first-line treatment of patients with AL amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged between 18 to 80 years
* Renal or other type biopsy was used to diagnose AL amyloidosis
* Understand and voluntarily sign an informed consent form
* ECOG score 0-3 points
* Adequate residual organ function

Exclusion Criteria:

* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Grade 3 sensory or grade 1 painful peripheral neuropathy
* Known hypersensitivity to bortezomib, boron or mannitol
* Cardiac syncope, uncompensated New York Heart Association (NYHA) Class 3 or 4 congestive heart failure
* Clinically overt multiple myeloma
* Pregnant or nursing women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from hospital，who were diagnosed AL amyloidosis by renal or other type biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hematologic response rate | 3 months
  Hematologic responses were evaluated according to the novel criteria of the International Society of Amyloidosis

SECONDARY OUTCOMES:
organ response rate | 12 months
  organ responses were evaluated according to the novel criteria of the International Society of Amyloidosis
Overall survival | From date of the start of treatment to date of death,up to 3 months
Progression free survival | From date of the start of treatment to date of disease progression,up to 3 months